CLINICAL TRIAL: NCT02839616
Title: Institutional Registry of Liver Transplantation
Acronym: IRLT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital El Cruce (Other)
Responsible Party: Principal Investigator, Liliana Paloma Rojas Saunero, Research fellow, Hospital El Cruce
Other Study IDs: 120716/1
Record Dates: First submitted 2016-07-15; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Liver Transplantation; Clinical Registry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: orthotopic liver transplantation

SUMMARY:
The Institutional Registry of Liver Transplantation is a system for data collection related to patients with liver disease who are possible candidates for liver transplantion. This tool was designed by a multidisciplinary team that includes hepatologists, surgeons, informatics and biostatisticians. It intends to collect the information from the clinical evaluation, physical examination, complementary diagnostic methods and laboratory data. The information is captured sistematically, following structured, standardized and monitored processess to ensure the quality of the data obtained.

The aim is to use the available technology to generate a complete database that can be used to answer research questions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for liver transplantation
* Patients who are followed by the Liver Transplantation Unit of Hospital El Cruce

Exclusion Criteria:

* Patients who deny to participate after the informed consent process.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic liver disease or acute liver failure who are candidates for liver transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Time to mortality | 5 years
  All patients are followed from the date of the inclusion to the registry, by periodic controls by the hepatologists and through telephones calls by the coordinator nurse, both before and after the transplantation.
  Every patient who dies during the 5 years of follow up will count as an event. Patients who are lost to follow up will be censored, in this case we will use the date of the last control or telephone call where he or she was alive.

SECONDARY OUTCOMES:
Time to retransplantation | 5 years
  We will considerate retransplantation as a competitive risk for death, calculating the time since the date of the transplant until the date of retransplantantion or not during the 5 years of follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Liliana P Rojas Saunero, MD, Principal Investigator — Hospital El Cruce
Locations (1):
- Hospital de Alta Complejidad El Cruce, Provincia Florencio Varela, Buenos Aires, Argentina

REFERENCES:
- [Background] Dickinson DM, Ellison MD, Webb RL. Data sources and structure. Am J Transplant. 2003;3 Suppl 4:13-28. doi: 10.1034/j.1600-6143.3.s4.3.x. No abstract available. PMID 12694047
- [Background] Leppke S, Leighton T, Zaun D, Chen SC, Skeans M, Israni AK, Snyder JJ, Kasiske BL. Scientific Registry of Transplant Recipients: collecting, analyzing, and reporting data on transplantation in the United States. Transplant Rev (Orlando). 2013 Apr;27(2):50-6. doi: 10.1016/j.trre.2013.01.002. Epub 2013 Mar 6. PMID 23481320
- [Background] Koller MT, van Delden C, Muller NJ, Baumann P, Lovis C, Marti HP, Fehr T, Binet I, De Geest S, Bucher HC, Meylan P, Pascual M, Steiger J. Design and methodology of the Swiss Transplant Cohort Study (STCS): a comprehensive prospective nationwide long-term follow-up cohort. Eur J Epidemiol. 2013 Apr;28(4):347-55. doi: 10.1007/s10654-012-9754-y. Epub 2013 Apr 2. PMID 23546766
- [Background] Schaubel DE, Dykstra DM, Murray S, Ashby VB, McCullough KP, Dickinson DM, Hulbert-Shearon TE, Webb RL, Wolfe RA. Analytical approaches for transplant research, 2004. Am J Transplant. 2005 Apr;5(4 Pt 2):950-7. doi: 10.1111/j.1600-6135.2005.00837.x. PMID 15760420